CLINICAL TRIAL: NCT00250874
Title: Phase I-II Study of Liposomal Doxorubicin (Myocet®), Docetaxel and Trastuzumab as First-Line Treatment of Patients With HER-2/Neu Positive Metastatic Breast Cancer
Brief Title: Myocet, Docetaxel & Trastuzumab as 1st Line Treatment of Patients With HER-2/Neu Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeneus Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myocet 008 (L017)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2005-11-08 (Estimated); Status verified 2005-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Doxorubicin; Docetaxel; Trastuzumab

INTERVENTIONS:
Drug: Liposomal Doxorubicin (Myocet), Docetaxel and Trastuzumab

SUMMARY:
To study the pharmacokinetic profile of the therapeutic schedule in order to demonstrate absence of negative interactions among the 3 drugs administered

DETAILED DESCRIPTION:
1. To assess the maximum tolerated dose (MTD) of Myocet at different dosages in combination with Taxotere at the fixed dose of 35 mg/m2 on day 2 and 9 every 21 days and weekly Herceptin as first line therapy in patients affected by HER-2/neu positive metastatic breast cancer
2. To enhance the proportion of complete remission
3. To allow the feasibility of the combination of Herceptin with both Myocet and Taxotere without an enhanced risk of cardiotoxicity

ELIGIBILITY:
Inclusion Criteria:

* HER-2/neu overexpression assessed by FISH test or with immunohistochemical methods: Dako(the result must be 3+ with dakotest); if the immunohistochemical test results 2+ it is needed a positive FISH test
* Female < 70yrs
* Histologically or cytologically proven breast cancer.
* Metastatic or locally advanced breast cancer (clinical stage: III-IV)
* Adequate hematological, hepatic, renal and cardiac function, the latter confirmed by echocardiography with FEVS ≥50%
* Prior adjuvant chemotherapy if doxorubicin total dose ≤300 mg/m2, epirubicin total dose ≤450 mg/m2

Exclusion Criteria:

* History of cardiopathy
* Severe hepatic and renal diseases
* Brain metastases as the only parameter of disease
* Contraindication to the use of corticosteroids as premedication
* Acute infectious diseases
* Insulin-dependent diabetes
* History of other cancers except for adequately treated basal cell skin cancer or in situ carcinoma of the cervix
* Concurrent treatment with any other cancer therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Professor Amadori, Principal Investigator — Ospedale Pietrantoni, Forli, Italy; Professor Gasparini, Principal Investigator — San Filippo Neri, Rome, Italy
Locations (1):
- Ospedale Pietrantoni, Forlì, Italy